CLINICAL TRIAL: NCT02812264
Title: Using an API to Commercialize an Evidence-Based Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coeus Health, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4R44DK103519-02 (NIH)
Record Dates: First submitted 2016-06-10; First posted 2016-06-24 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Weight Loss; Health Behavior
MeSH Terms: conditions — Weight Loss; Health Behavior | interventions — Fitness Trackers; Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will not know which arm they have been randomized to. Additionally, the investigators will be blinded to participant assignment. Randomization will be completed by the program manager.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- API App (Experimental): use of API weight loss mobile application for 12 months, plus fitness tracker and scale.
  Interventions: Behavioral: API App; Behavioral: fitness tracker; Behavioral: scale
- Attention Control (Active Comparator): use of non-API app for weight loss over 12 months, plus fitness tracker and scale.
  Interventions: Behavioral: Non-API App; Behavioral: fitness tracker; Behavioral: scale

INTERVENTIONS:
Behavioral: API App — Mobile application that uses API technology to deliver evidence-based weight loss intervention. Includes syncing with wearable fitness tracker and scale
  Arms: API App
Behavioral: Non-API App — Mobile application that does not use API technology to deliver evidence-based weight loss intervention. Includes syncing with wearable fitness tracker and scale.
  Arms: Attention Control
Behavioral: fitness tracker — fitness tracker to monitor physical activity and sleep patterns that is connected to transfer data to app
  Other Names: wearable
Behavioral: scale — Connected scale that will transfer weight information to app
  Other Names: weight

SUMMARY:
This study will test the effectiveness of a mobile application that uses an Application Program Interface (API) to distribute evidence-based weight loss interventions. Half of the participants will receive this API-based application, and the other half of the participants will use a non API-based application.

DETAILED DESCRIPTION:
The purpose of this study is to test a weight loss app that uses an API to disseminate an evidence-based weight loss intervention. The investigators hypothesize that, over the course of 12 months, participants using the Leaner app will have lost more weight than those in the attention control group.

Participants (n=206) will be randomly assigned to use either the intervention app (intervention arm; n=103) or a weight loss app of their choosing (attention control arm; n=103) for 12 months. Assessments will take place at baseline, and 3, 6, and 12 months.

Statistical analysis: A linear mixed modeling approach will be used to test the hypothesis. Observed weight vs. time plots will be analyzed for all participants to discern general trends in weight change. The model will include an intervention effect, a time effect, an intervention by time interaction, and a random intercept.

In exploratory analysis, investigators will examine weight change across subgroups of interest; investigators will add the subgroup variable and its interaction with the intervention indicator to the primary model. All analyses will be evaluated at the 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 21-65 years old
* BMI between 25-40 kg/m2
* ownership and use of an Android smartphone during past 6 months with no plans to change phone/service during study
* consent for research team to monitor app utilization

Exclusion Criteria:

* use of weight loss medication
* prior or planned bariatric surgery
* psychiatric hospitalization in past 12 months
* pregnancy, nursing, or planned pregnancy during the study
* history of cardiovascular disease (CVD) event
* self-reported history of an eating disorder
* use of medication for diabetes mellitus
* mobility restrictions for which exercise is contraindicated
* history of a condition (e.g., lithium, steroids, anti-psychotics) that would affect weight measurement, for which weight loss is contraindicated
* current participation in another weight treatment study and/or recent weight loss >10%
* investigator discretion for safety reasons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Weight change | up to 12 months
  Change in body weight over course of study

SECONDARY OUTCOMES:
Weight Change - 3 months | up to 3 months
  Initial weight change
Weight Change - 6 months | up to 6 months
  mid-point weight change
Automated Self-Administered 24-hour Dietary recall (ASA-24) | baseline, 3-, 6-, 12-months
  Dietary patterns/24-hour dietary recall
Physical Activity | baseline, 3-, 6-, 12-months
  Paffenbarger survey to capture physical activity patterns. Assesses self-report leisure time physical activity and weekly kilocalorie expenditure.
Blood Pressure | baseline, 3-, 6-, 12-months
  Using a blood pressure cuff, measured three times at 1-minute intervals after 5 minutes of quiet sitting. Average of final two measurements is used.
Fasting Lipid Profile | baseline, 3-, 6-, 12-months
  finger stick blood samples will be collected, following an overnight fast, to analyze fasting lipid profile. Samples will be analyzed using the Cholestech LDX
Plasma Glucose | baseline, 3-, 6-, 12-months
  finger stick blood samples will be collected, following an overnight fast, to analyze plasma glucose. Samples will be analyzed using the Cholestech LDX
High Sensitivity C-Reactive Protein | baseline, 3-, 6-, 12-months
  finger stick blood samples will be collected, following an overnight fast, to analyze high sensitivity c-reactive protein. Samples will be analyzed using the Cholestech LDX
Patient Health Questionnaire (PHQ) 9 | baseline, 3-, 6-, 12-months
  Nine-item self-report assessment of depression severity.
Body Shape Questionnaire (BSQ) | baseline, 3-, 6-, 12-months
  8-item self-report questionnaire about concern with body shape.
Mizes Anorectic Cognitions Questionnaire - Revised (MAC-R) | baseline, 3-, 6-, 12-months
  24-item self-report measure of disordered eating cognitions.
Questionnaire of Eating and Weight Patterns | baseline, 3-, 6-, 12-months
  Eight-item self-report measure of binge eating behaviors.
Medical Outcomes Survey: Social Support | baseline, 3-, 6-, 12-months
  19-item self-report assessment of social support.
EuroQOL Health Related Quality of Life Scale | baseline, 3-, 6-, 12-months
  16-item self-report assessment of health related quality of life.
The Health and Work Performance Questionnaire (HPQ) | baseline, 3-, 6-, 12-months
  Presenteeism/Absenteeism items from the self-report HPQ.
App engagement | through study completion, an average of 1 year
  Using technology on smart phones, we will monitor participants' app usage throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Coeus Health Offices, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided